CLINICAL TRIAL: NCT04516174
Title: Effect of Transversus Abdominis Plane Block Combined With Dexmedetomidine Infusion on the Prognosis in Elderly Patients Undergoing Abdominal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Vice Professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: wys20200731
Record Dates: First submitted 2020-08-11; First posted 2020-08-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Colorectal Neoplasms; Aged
Keywords: Delirium; Pain, Postoperative; Dexmedetomidine; Transversus abdominis plane block
MeSH Terms: conditions — Colorectal Neoplasms; Delirium; Pain, Postoperative | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dex+TAPB group (Experimental): Patients in Dex+TAPB group will receive the bilateral transversus abdominis plane block with 0.25% ropivacaine 20ml each side before anesthesia and combined with continuous infusion of dexmedetomidine during operation.
  Interventions: Procedure: Transversus abdominis plane block using ropivacaine; Drug: Dexmedetomidine
- Control group (Placebo Comparator): Patients in control group will receive the bilateral transversus abdominis plane block with saline 20ml each side before anesthesia and don't receive the infusion of dexmedetomidine during operation.
  Interventions: Procedure: Transversus abdominis plane block using saline; Drug: Saline

INTERVENTIONS:
Procedure: Transversus abdominis plane block using ropivacaine — Before anesthesia, the ultrasound-guided bilateral transversus abdominis plane block using 0.25% ropivacaine was perdormed by anesthesiologist who is not involved in intraoperative management and postoperative follow-up and evaluate the effect after the block completed.
  Arms: Dex+TAPB group
Drug: Dexmedetomidine — After finished the transversus abdominis plane block, then perform tracheal intubation and start the infusion of dexmedetomidine.
  Arms: Dex+TAPB group
Procedure: Transversus abdominis plane block using saline — Before anesthesia, the ultrasound-guided bilateral transversus abdominis plane block using saline was perdormed by anesthesiologist who is not involved in intraoperative management and postoperative follow-up and evaluate the effect after the block completed.
  Arms: Control group
Drug: Saline — After finished the transversus abdominis plane block, then perform tracheal intubation and start the infusion of saline, dosage and infusion method of saline are consistent with dexmedetomidine.
  Arms: Control group

SUMMARY:
To compare the prognosis of elderly patients undergoing radical resection of colorectal cancer treated with general anesthesia and general anesthesia combined with transversus abdominis plane block and continuous infusion of dexmedetomidine. The incidence of postoperative delirium, postoperative acute pain moderately to severely and poor postoperative recovery were composite endpoints to determine the prognosis of patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 65-80 years,regardless of gender
* American Society of Anesthesiologists physical status I-III
* Undergoing elective radical resection of colorectal cancer
* Sign informed consent

Exclusion Criteria:

* Could not cooperate to complete the pain VAS evaluation
* Could not cooperate to complete the cognitive function assessment

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2020-09-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
The prognosis of aged patients | Postoperative 72 hours
  The incidence of postoperative delirium, postoperative acute pain moderately to severely and poor postoperative recovery were composite endpoints to determine the prognosis of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tian Tan Hospital, Beijing, China